CLINICAL TRIAL: NCT02427984
Title: Early Diagnosis of Pending Failures of Total Hip Arthroplasty With Hard to Hard Bearings
Brief Title: Pending Failure in Hard-hard Total Hip Arthroplasty
Acronym: PF
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Susanna Stea, M.sc., Istituto Ortopedico Rizzoli
Other Study IDs: IORizzoli
Record Dates: First submitted 2015-02-19; First posted 2015-04-28 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Infection and Inflammatory Reaction
Keywords: Internal Left Hip Prosthesis; Internal Right Hip Prosthesis
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, synovial fluid, urines, periprosthetic tissues, at -80°C
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Metal on Metal (MoM): Patients wearing MoM hip prosthesis
  Interventions: Other: Metal ions dosage and evaluation of local/systemic reaction
- Ceramic on Ceramic (CoC): Patients wearing CoC hip prosthesis
  Interventions: Other: Noise registration and metal ions determination
- Controls: Patients free from hip devices
  Interventions: Other: Metal ions dosage, evaluation of local/systemic reaction, noise registration

INTERVENTIONS:
Other: Metal ions dosage and evaluation of local/systemic reaction — Dosage of Chromium and Cobalt on several biological matrices deriving from each patients.
  Determination of local/systemic reaction
  Groups: Metal on Metal (MoM)
Other: Noise registration and metal ions determination — Dosage of Vanadium and Titanium on several biological matrices deriving from each patients.
  Determination of range of noise
  Groups: Ceramic on Ceramic (CoC)
Other: Metal ions dosage, evaluation of local/systemic reaction, noise registration — Dosage of Chromium, Cobalt, Vanadium and Titanium on several biological matrices deriving from each patients.
  Determination of local/systemic reaction
  Other Names: Controls comparison for variables considered
  Groups: Controls

SUMMARY:
During last 6 years approximately 10.000 ceramic balls and 5.000 ceramic liners have been implanted in the region Emilia-Romagna in Italy (4 million Every single year approximately 60.000 hip prostheses are implanted in Italy. Quality of life of patients after surgery is very good, as widely demonstrated in the literature. On the basis of data produced by the only complete hip register in Italy that is run in our Lab (RIPO, Register of Orthopedic Implants in the Region Emilia-Romagna) survival rate of primary total hip prosthesis is 95.6% at 9 years. Reasons for revision are mainly aseptic loosening of one or both components (40% of the total) and dislocation (26%), being the latter much more frequent in the first two years. Less frequently revision is due to sepsis (7% of the total),bone fracture (11%), prosthesis fracture (3%) or pain (3%). Revision is relates, among the others, to prosthesis-related factors, such as fixation to bone and articular coupling. In our experience, during the last ten years 32% of implants had both articular component in ceramic , 34% had metal head and plastic liner, 24% ceramic head and plastic liner, 10% both components in metal.

Each solution has strengths and weakness and they have been identified and clinically applied in order to overcome step by step limitations observed in the previous one. The most recent are the hard-on-hard bearings, that is ceramic on ceramic and metal on metal. These two solutions, beside very promising results on wear resistance, show some peculiar failures: respectively fracture of the ceramic component and hypersensitivity induced by metal ions.

Aim of research proposal is to investigate two uncommon and less investigated early symptoms of failure:

* 'noising hip' in ceramic on ceramic total hip arthroplasty
* pain without radiographic signs of loosening in metal on metal total hip arthroplasty These two situations are extremely relevant, as they prelude to a failure of the prosthesis. If clearly identified they could represent a powerful tool in early diagnosis of pending failure To reach this goal our patients wearing hard-on-hard total hip arthroplasty, suffering for described symptoms will undergone a specific diagnostic procedure.

The first group will be studied through CT scan of the patients to evaluate impingement or instability of the prosthesis, and a needle aspiration for synovial fluid. The fluid will be examined to identify ceramic wear debris, according to a method of separation and analysis in scanning electron microscopy that was set in our Lab.

Sound will be recorded by means of a wearable sensor set capable of recording the articular noise produced during level walking. This instrumentation will be coupled to motion analysis technology.

This would make possible a diagnostic approach able to correlate the involved factors to clinical occurrences, on the basis of the recorded frequencies.

-Second group will be studied through the dosage of circulating ions, deriving from the articular surfaces and through the histological classification of vasculitis in periimplant tissues. There is increasing evidence, indeed that locale release of submicron particles worn out from articular surfaces can release metal ions (mainly Chromium and Cobalt) responsible for lymphocyte local infiltration. In particular CD20 positive B lymphocyte and CD3 positive T lymphocyte and sometimes CD68 positive plasma cells are present. The cells could justify the development of pseudotumors in metal-on metal hip prosthesis.

Data collected from patients matched to in vitro results will allow us to to avoid or at least propose a more appropriate timing for revision surgery.

DETAILED DESCRIPTION:
Every single year approximately 60.000 hip prostheses are implanted in Italy. Quality of life of patients after surgery is very good, as widely demonstrated in clinical experience and in the literature. On the basis of data produced by the only complete hip register in Italy, that is run in our Lab (RIPO, Register of Orthopedic Implants in the Region Emilia-Romagna http://ripo.cineca.it) survival rate of primary total hip prosthesis is 95.6% at 9 years. Reasons for revision are mainly aseptic loosening of one or both components (40% of the total) and dislocation (26%), being the latter much more frequent in the first two years. Less frequently revision is due to sepsis (7% of the total),bone fracture (11%), prosthesis fracture (3%) or pain (3%).

Revision can be related, among the others, to prosthesis-linked factors, such as fixation to bone and articular coupling.

In the experience of RIPO, during the last ten years 32% of implants had both articular component in ceramic, 34% had metal head and plastic liner, 24% ceramic head and plastic liner, 10% both components in metal.

Each solution has strengths and weakness and they have been identified and clinically applied in order to overcome step by step limitations observed in the previous one.

Alumina ceramic-on-ceramic (COC) bearings have been shown to produce substantially less wear debris than traditional metal/ceramic on polyethylene bearings. In addition, the alumina ceramic material itself is essentially bioinert in both bulk and particulate form . Unlike metal-on-metal bearings (MOM), this bearing couple does not release metal ions into the body either from the articulation or from breakdown of wear debris. Weakness of ceramic-on-ceramic bearings are represented by brittleness of the material. Ceramic can fracture, even in very few cases, due to trauma or to malpositioning. Beside this occurrence of noise during gait of patients can be extremely disturbing for patient itself, leading to request of revision. These two solutions represent more recent proposal that technology suggested to overcome problem of wear.

Hard components on plastic has the unsolved problem of wear debris, leading to osteolysis and consequent failure of he im plant. The problem has only partially solved by the introduction of cross linked polyethylene, aimed to improve tribological behaviour of the plastic.

Rizzoli Institute is the only public mono-specialistic research hospital in Italy. Nearly 500 hip prosthesis revisions are performed here every year in the structure. Due to its high specialization difficult cases from all the country are treated here, not on ly when anatomy of the patient is damaged (dislocation of the hip, post traumatic arthritis) but .even more frequently when failure of the implant occurred.

Aim of research proposal is to investigate two uncommon and less investigated early symptoms of failure:

* 'noising hip' in ceramic on ceramic total hip arthroplasty
* pain in metal on metal total hip arthroplasty Even if not numerically so important, these two situations are extremely relevant, as they prelude to a failure of the prosthesis. If clearly identified they could represent a powerful tool in early diagnosis of pending failure.

The first point will be studied through CT scan of the patients to evaluate impingement or instability of the prosthesis, and a needle aspiration for synovial fluid. The fluid will be examined to identify ceramic wear debris, according to a method of separation and analysis in scanning electron microscopy that was set in our Lab.

Sound will be recorded by means of a wearable sensor set capable of recording the articular noise produced during level walking. This instrumentation will be coupled to motion analysis technology, so as to provide a temporal correlation between the recorded noise and the gait cycle. It will be developed in the first phase of the project. In parallel surface analyses will be conducted on retrievals that are stored in the Lab since 2000, in one of the biggest retrieval study ever conducted in our country. Type of damage, surface roughness of both ceramic components will be analysed and compared to clinical data.

Finally the study will be completed in vitro, using an hip simulator, to reproduce the possible clinical scenarios leading to hip noise, record, and analyse it in a reproducible and robust manner. This would make possible a diagnostic approach able to correlate the involved factors to clinical occurrences, on the basis of the recorded frequencies. Second point will be studied through the dosage of circulating ions, deriving from the articular surfaces and through the histological classification of vasculitis in periimplant tissues. There is increasing evidence, indeed that locale release of submicron particles worn out from articular surfaces can release metal ions (mainly Chromium and Cobalt) responsible for lymphocyte local infiltration. In particular cluster of differentiation antigen 20 (CD20) positive B lymphocyte and cluster of differentiation 3 (CD3) positive T lymphocyte and sometimes cluster of differentiation antigen 68 (CD68) positive plasma cells are present. The cells could indicate a specific phlogistic condition responsible for pain and eventually subsequent revision.

Data collected on studied population will allow a better understanding of the two phenomena and possibly will suggest new therapeutic approaches to the problems.

ELIGIBILITY:
Inclusion Criteria:

* Patient waiting for primary total hip arthroplasty (THA)
* Patients MoM and CoC referring to our ward
* Informed consent approved
* Questionnaire on habits filled

Exclusion Criteria:

* Sepsis or suspected sepsis
* Patients exposed to other font of metals

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients (no septic) afferent to our ward and wearing hip prosthesis MoM or CoC. A group of control patients, waiting for primary total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2012-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Toni, MD, Study Director — Istituto Ortopedico Rizzoli
Locations (1):
- Laboratorio Tecnologia Medica, Bologna, Italy, Italy

REFERENCES:
- [Result] Beraudi A, Stea S, De Pasquale D, Bordini B, Catalani S, Apostoli P, Toni A. Metal ion release: also a concern for ceramic-on-ceramic couplings? Hip Int. 2014 Jul-Aug;24(4):321-6. doi: 10.5301/hipint.5000132. Epub 2014 Mar 24. PMID 24817392
- [Result] Beraudi A, Catalani S, Montesi M, Stea S, Sudanese A, Apostoli P, Toni A. Detection of cobalt in synovial fluid from metal-on-metal hip prosthesis: correlation with the ion haematic level. Biomarkers. 2013 Dec;18(8):699-705. doi: 10.3109/1354750X.2013.846413. Epub 2013 Oct 17. PMID 24134776
- [Result] Catalani S, Stea S, Beraudi A, Gilberti ME, Bordini B, Toni A, Apostoli P. Vanadium release in whole blood, serum and urine of patients implanted with a titanium alloy hip prosthesis. Clin Toxicol (Phila). 2013 Aug;51(7):550-6. doi: 10.3109/15563650.2013.818682. Epub 2013 Jul 11. PMID 23845123
- [Result] De Pasquale D, Stea S, Beraudi A, Montesi M, Squarzoni S, Toni A. Ceramic debris in hip prosthesis: correlation between synovial fluid and joint capsule. J Arthroplasty. 2013 May;28(5):838-41. doi: 10.1016/j.arth.2013.01.019. Epub 2013 Mar 13. PMID 23489725

RESULTS

PARTICIPANT FLOW:
Groups:
- Metal on Metal (MoM): All the patients of our Division with MoM THA
- Ceramic on Ceramic (CoC): All the patients of our Division with CoC THA
Period: Overall Study
Arm/Group | Metal on Metal (MoM) | Controls | Ceramic on Ceramic (CoC)
Started | 53 | 45 | 50
Completed | 40 | 40 | 32
Not Completed | 13 | 5 | 18
Not completed — Lost to Follow-up | 13 | 5 | 18

BASELINE CHARACTERISTICS:
Groups:
- Controls: All the patients of our Division for primary THA
- Total: Total of all reporting groups
Arm/Group | Metal on Metal (MoM) | Controls | Ceramic on Ceramic (CoC) | Total
Number analyzed (Participants) | 40 | 40 | 32 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 20 | 20 | 12 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 20 | 65
  Male | 20 | 15 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Chromium and Cobalt Ion Levels Above 7ug/l
Description: Measured by Inductively coupled plasma mass spectrometry (ICP-MS), equipped with dynamic cell reaction (ELAN DRC II) and expressed in micrograms/liter.
  Will be counted the number of patients with level os metals above 7micrograms/liter
  This outcome is valuable only for MoM arm and Control arm (as comparison), because CoC arm patients don't wear device releasing this kind of metals.
Time Frame: 3 years
Population: the population was evaluated as number of patients with ions level above 7ug/l (attention limit)
Measure: Number; unit: participants above limit
Arm/Group | Metal on Metal (MoM) | Control
Number analyzed (Participants) | 40 | 40
participants above limit | 14 | 0

2. Primary Outcome: Duration of Articular Noise Produced During Level Walking
Description: Measured by fast Fourier transform (FFT) expressed in duration (milliseconds)
  This outcome is valuable only for CoC arm and MoM arm, because Control arm patients don't wear prosthesis (no noise)
Time Frame: 3 years
Measure: Mean (Full Range); unit: milliseconds
Arm/Group | Ceramic on Ceramic (CoC) | Metal on Metal (MoM)
Number analyzed (Participants) | 32 | 40
milliseconds | 174 [40 to 300] | 40 [40 to 300]

3. Primary Outcome: Frequency of Articular Noise Produced During Level Walking
Description: Measured by fast Fourier transform (FFT) expressed in frequency (Hz) This outcome is valuable only for CoC arm and MoM arm, because Control arm patients don't wear prosthesis (no noise)
Time Frame: 3 years
Measure: Mean (Full Range); unit: Hz
Arm/Group | Ceramic on Ceramic (CoC) | Metal on Metal (MoM)
Number analyzed (Participants) | 32 | 40
Hz | 910 [100 to 1500] | 100 [100 to 1500]

4. Primary Outcome: Amplitude of Articular Noise Produced During Level Walking
Description: Measured by fast Fourier transform (FFT) expressed in amplitude (decibel) This outcome is valuable only for CoC arm and MoM arm, because Control arm patients don't wear prosthesis (no noise)
Time Frame: 3 years
Measure: Mean (Full Range); unit: decibel
Arm/Group | Ceramic on Ceramic (CoC) | Metal on Metal (MoM)
Number analyzed (Participants) | 32 | 40
decibel | -20 [-38 to -2] | -38 [-38 to -2]

5. Secondary Outcome: Number of Participants Who Scored Positive for ALVAL
Description: Histological score defined by the valuation of staining It was possible to valuate this outcome only for 29 out of 40 patients MoM (due to the availability of periprosthetic tissues).
  The arms CoC and controls were not studied for this issue because ALVAL could occur only in presence of Metals
Time Frame: 3 years
Population: positive for ALVAL is +, negative for ALVAL is -
Measure: Number; unit: participants
Arm/Group | Metal on Metal (MoM)
Number analyzed (Participants) | 29
participants | 15

ADVERSE EVENTS:
Arm/Group | Metal on Metal (MoM) | Ceramic on Ceramic (CoC) | Controls
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/32 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/32 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No